CLINICAL TRIAL: NCT02315287
Title: Comparison of Therapeutic Efficacy Between Lobeglitazone and Pioglitazone as Initial Triple Therapy With Metformin and Sitagliptin in Drug-naïve Type 2 Diabetic Patients
Brief Title: Comparison of Lobeglitazone With Pioglitazone as Initial Triple Therapy for Diabetes Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lobe vs. Pio
Record Dates: First submitted 2014-09-11; First posted 2014-12-11 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
Keywords: Triple combination; Metformin; Sitagliptin; Pioglitazone; Lobeglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; lobeglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin, Sitagliptin, Pioglitazone (Active Comparator): Thiazolidinedione
  Interventions: Drug: Pioglitazone
- Metformin, Sitagliptin, Lobeglitazone (Active Comparator): Thiazolidinedione
  Interventions: Drug: Lobeglitazone

INTERVENTIONS:
Drug: Pioglitazone — Comparison of two different thiazolidinediones
  Other Names: Actos
  Arms: Metformin, Sitagliptin, Pioglitazone
Drug: Lobeglitazone — Comparison of two different thiazolidinediones
  Other Names: Duvie
  Arms: Metformin, Sitagliptin, Lobeglitazone

SUMMARY:
Triple combination of metformin, DPP4 inhibitor and Thiazolidinedione would be a good option in the treatment of drug-naïve Korean type 2 diabetic patients. Newly developed thiazolidinedione, Lobeglitazone would be not inferior to Pioglitazone.

DETAILED DESCRIPTION:
Thiazolidionedione, a PPARgamma agonist, is an strong insulin sensitizer. It has shown that durable glucose lowering effect and beta cell preservation. It is an important treatment option in patients with type 2 diabetes.

It has been well established that inhibition of dipeptidyl peptidase-4 (DPP-4) reduces blood glucose levels in both fasting and postprandial states, and preserves pancreatic β-cell function in patients with type 2 diabetes. The mechanism of action of DPP-4 inhibitors is to increase levels of active incretin, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), which stimulate insulin secretion as well as insulin biosynthesis while inhibiting glucagon release from pancreatic islets.

DPP4 inhibitors also have better safety and tolerability profiles (e.g., weight neutrality and less hypoglycemia) compared to other hypoglycemic agents. When considering combination therapy with DPP-4 inhibitors, metformin is the most commonly used agent which has been shown to be effective and well tolerated from previous studies. Besides the glucose lowering effect by reducing hepatic glucose output and improving insulin resistance, metformin without inhibiting DPP-4 activity,also increases active GLP-1 concentrations by 1.5- to 2-fold following an oral glucose load in obese, nondiabetic subjects. Accordingly, this effect of metformin may provide a unique benefit when combined with DPP-4 inhibitors through a substantial enhancement of the incretin axis, which provides effective and potentially additive glycemic improvement.

Because of its favorable pharmacological properties, combination of a DPP-4 inhibitor, metformin, and thiazolidinedione has been increasingly used to achieve rapid glycemic goal with low risk of hypoglycemia and no weight gain, and to delay the need for subsequent regimen changes. DPP-4 inhibitors block DPP-4 enzyme and preserve endogenous incretins whereas metformin increases the active form of GLP-1, both of which may enhance the secretory function of pancreas. However, the response to DPP-4 inhibitors and metformin combination therapy may be different in individuals according to their pancreatic function and insulin resistance status. In fact, previous studies with DPP-4 inhibitors showed different potency in glycemic controls depending on various patient characteristics including severity of diabetes and the use of other antidiabetic drug.Consequently, it would be clinically important to investigate effect of this triple combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 13.0 %
* No treatment with insulin or oral agents for 6 months
* 20 ≤ Age < 80 years

Exclusion Criteria:

* Contraindication to sitagliptin or metformin or thiazolidinedione
* Pregnant or breast feeding women
* Type 1 diabetes, gestational diabetes, or secondary forms of diabetes
* Not appropriate for oral antidiabetic agent
* Medication which affect glycemic control
* Disease which affect efficacy and safety of drugs
* Any major illness (Liver disease, Renal failure, Heart disease, Cancer, etc)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c | 5 and 12 months
  Comparison of therapeutic efficacy of two thiazolidinediones (Piogitazone vs. Lobeglitazone) in drug-naïve Korean type 2 diabetic patients

SECONDARY OUTCOMES:
Beta-cell function | 12 months
  Changes of beta-cell function after 12 months treatment of triple combination
Insulin resistance | 12 months
  Changes of insulin resistance after 12 months treatment of triple combination
HbA1c < 7.0% | 5 and 12 months
  Comparision of glycemic control
HbA1c =< 6.5% | 5 and 12 months
  Comparision of glycemic control
FBS and PP2 | 5 and 12 months
  Comparision of glycemic control
microalbumin to creatinine ratio | 5 and 12 months
  Comparision of albumiuria

OTHER OUTCOMES:
Hypoglycemia | 12 months
  Incidence of hypoglycemia in triple combination treatment
Body weight | 12 months
  Changes of weight after 12months treatment of triple combination

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea